# UNIVERSITY OF MICHIGAN CONSENT TO BE PART OF A RESEARCH STUDY

#### 1. KEY INFORMATION ABOUT THE RESEARCHERS AND THIS STUDY

Study title: Precision Antibiotic Dosing for Appendectomy (PANDA Study)

Company or agency sponsoring the study: Agency for Healthcare Research and Quality

Names, degrees, and affiliations of the principal investigator and study coordinator (if applicable):

Principal Investigator: Manjunath (Amit) Pai, PharmD, Clinical Pharmacy, University of Michigan

#### 1.1 Key Study Information

You may be eligible to take part in a research study. This form contains important information that will help you decide whether to join the study. Take the time to carefully review this information. You should talk to the researchers about the study and ask them any questions you have. You may also wish to talk to others such as your family, friends, or other doctors about joining this study. If you decide to join the study, you will be asked to sign this form before you can start study-related activities. Before you do, be sure you understand what the research study is about.

A research study is different from the regular medical care you receive from your doctor. Research studies hope to make discoveries and learn new information about diseases and how to treat them. You should consider the reasons why you might want to join a research study or why it is not the best decision for you at this time.

Research studies do not always offer the possibility of treating your disease or condition. Research studies also have different kinds of risks and risk levels, depending on the type of the study. You may also need to think about other requirements for being in the study. For example, some studies require you to travel to scheduled visits at the study site in Ann Arbor or elsewhere. This may require you to arrange travel, change work schedules, find childcare, or make other plans. In your decision to participate in this study, consider all these matters carefully.

This research is studying a drug called cefoxitin already approved by the Food and Drug Administration (FDA) to reduce the risk of infection after surgery to remove an appendix. Researchers are studying a large group of people to continue to learn how best to dose antibiotics. This research will compare the current standard treatment which is a single dose prior to surgery to a new method that includes adding another dose of cefoxitin within 30 minutes of starting the surgery. If you participate in this study, we will collect three blood samples, two fat samples, and a sample of your appendix collected during the surgery. We will measure drug concentrations in these samples to compare the standard dosing method to our new method. Your health-related information will also be collected for this research study.

This study involves a process called randomization. This means whether or not you receive the additional dose of cefoxitin in the study is not chosen by you or the researcher. The study design divides study participants into separate groups, based on chance (like the flip of a coin), to compare current standard dosing to a new dosing method. If you decide to be in the study, you need to be comfortable not knowing which study group you will be in.

There can be risks associated with joining any research study. The type of risk may impact whether you decide to join the study. For this study, some of these risks may include a loss of confidentiality or discomfort from sample collection sites. More detailed information will be provided later in this document.

| IRBMED standard informed consent template<br>(working version) |
|----------------------------------------------------------------|
| Approved 4/10/2024 |
| Blue box instructions revised 8/21/2024 |
| DO NOT REMOVE THIS FIELD—IRBMED USE ONLY |

Consent Subtitle: \_\_\_Aim 3\_\_\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_\_

This study may not offer any benefit to you now but may benefit others in the future by helping to decide whether an addition dose of this antibiotic can reduce the risk of infection after surgery. More information will be provided later in this document.

We expect the amount of time you will participate in the study will be no longer than the time spent in the operating room.

You can decide not to be in this study. Alternatives to joining this study include receiving the standard of care.

Even if you decide to join the study now, you are free to leave at any time if you change your mind.

More information about this study continues in Section 2 of this document.

#### 2. PURPOSE OF THIS STUDY

#### 2.1 Study purpose:

Surgical site infection (SSI) is a very common healthcare-associated infection occurring in patients undergoing appendectomy. We are studying whether adding a second dose of the antibiotic cefoxitin during surgery can improve concentrations that prevent SSI.

#### 3. WHO MAY PARTICIPATE IN THE STUDY

Taking part in this study is completely **voluntary**. You do not have to participate if you don't want to. You may also leave the study at any time. If you leave the study before it is finished, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled.

#### 3.1 Who can take part in this study?

Any adult, age 18 and older, who is scheduled for an appendectomy can take part in this study

#### 3.2 How many people are expected to take part in this study?

46 total subjects are expected to participate in this study

#### 4. INFORMATION ABOUT STUDY PARTICIPATION

#### 4.1 What will happen to me in this study?

You are scheduled to undergo appendectomy surgery. During the surgery, three (approximately 3 mL or under teaspoon each) blood collections will occur at the following time points: within 30 to 60 minutes before the start of the surgery (incision is when they cut through skin), at surgical incision, and at the end of surgery. Two subcutaneous fat samples (0.4-1 gram each or a medium-sized blueberry) will also be collected on surgical incision and around the time of surgical closure. We will also take a sample of your appendix once it has been removed from your body. You have a one-in-two chance of receiving the standard antibiotic dose or the standard antibiotic dose plus an additional dose of cefoxitin.

We would also like your permission to keep some of your tissues and medical information collected in the main study, so that we may study it in future research. The future research may be similar to this study or may be completely different.

You can take part in the main study even if you decide not to let us keep your blood, fat, and medical information for future research.

IRBMED standard informed consent template
(working version)

Approved 4/10/2024
Blue box instructions revised 8/21/2024
DO NOT REMOVE THIS FIELD—IRBMED USE ONLY

Consent Subtitle: \_\_\_Aim 3\_\_\_\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_\_

#### 4.2 How much of my time will be needed to take part in this study?

We will be taking samples during and shortly after your procedure. As the samples are small and will be taken by the surgeons or operative staff, that will not add any time to the surgery.

#### 4.3 When will my participation in the study be over?

Your active participation in the study is completed once we have obtained the necessary samples. We will collect information from your medical records that relate to your surgery and recovery from this procedure. We anticipate your participation will be complete with 1 year. The entire study is expected to last approximately 5 years.

#### 5. INFORMATION ABOUT STUDY RISKS AND BENEFITS

### 5.1 What risks will I face by taking part in the study? What will the researchers do to protect me against these risks?

During your surgery, we will be taking blood, fat, and appendix samples from you. We anticipate no risks due to the small amounts we will be collecting. There is a rare chance of discomfort from the collection sites. To decrease any discomfort, we will be collecting blood through existing ports that have been placed for your surgery. Fat samples will be taken from areas of incision based on your surgery.

If you are randomized to the cefoxitin dosing group, you will get a drug and dose that is commonly used in surgery. The additional risk of this extra dose is not known.

Additionally, there may be a risk involving loss of confidentiality or privacy. For example, if individuals outside this study were to discover that you were a participant in this research, or if any collected identifiable genetic or health information were disclosed to unauthorized persons, there is a risk of discrimination by employers or insurance providers. The researchers have adopted privacy and confidentiality procedures to help prevent such disclosures. See Section 9 of this document for more information on how the study team will protect your confidentiality and privacy.

As with any research study, there may be additional risks that are unknown or unexpected.

Keep in mind, as well, that the committee (IRBMED) that reviews this study does not review risks associated with procedures that are conducted as part of your regular medical care and are not part of the research, including those marked "[Not research]" in section 4.1, above. Risks associated with your regular medical treatment should be discussed with your regular doctor.

#### 5.2 What happens if I get hurt, become sick, or have other problems as a result of this research?

The researchers have taken steps to minimize the risks of this study. Even so, you may still have problems or side effects, even when the researchers are careful to avoid them. Please tell the researchers listed in Section 10 about any injuries, side effects, or other problems that you have during this study. You should also tell your regular doctors or any other provider or hospital you visit.

#### 5.3 If I take part in this study, can I also participate in other studies?

Being in more than one research study at the same time, or even at different times, may increase the risks to you. It may also affect the results of the studies. You should not take part in more than one study without approval from the researchers involved in each study.

| | IRBMED standard informed consent template (working version) |
|---|-------------------------------------------------------------|
| | Approved 4/10/2024 |
| | Blue box instructions revised 8/21/2024 |
| ı | DO NOT REMOVE THIS FIELD—IRBMED USE ONLY |

Consent Subtitle: \_\_\_Aim 3\_\_\_\_\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_\_\_

#### 5.4 How could I benefit if I take part in this study? How could others benefit?

You may not receive any personal benefits from being in this study. However, others may benefit from the knowledge gained from this study.

# 5.5 Will the researchers tell me if they learn of new information that could change my willingness to stay in this study?

Yes, the researchers will tell you if they learn of important new information that may change your willingness to stay in this study. If new information is provided to you after you have joined the study, it is possible that you may be asked to sign a new consent form that includes the new information.

#### 6. ALTERNATIVES TO PARTICIPATING IN THE STUDY

#### 6.1 If I decide not to take part in this study, what other options do I have?

Participating in this study is completely voluntary, your only alternative is not to participate, in which case, there are no penalties.

#### 7. ENDING THE STUDY

#### 7.1 If I want to stop participating in the study, what should I do?

You are free to leave the study at any time. If you leave the study before it is finished, there will be no penalty to you. You will not lose any benefits to which you may otherwise be entitled. If you choose to tell the researchers why you are leaving the study, your reasons for leaving may be kept as part of the study record. If you decide to leave the study before it is finished, please tell one of the persons listed in Section 10 "Contact Information".

#### 7.2 Could there be any harm to me if I decide to leave the study before it is finished?

You are free to end your participation partially or completely in the study. An example of partially ending your participation would be to discontinue receiving study intervention, while still allowing continuation of study follow-up procedures.

Please note that any information collected before you withdraw will be kept and used to complete the research.

Please note that even if you withdraw consent for further follow-up or contacts, if the study doctor becomes aware of additional safety information this will be reported to the sponsor to comply with legal or regulatory requirements.

#### 7.3 Could the researchers take me out of the study even if I want to continue to participate?

Yes. There are many reasons why the researchers may need to end your participation in the study. Some examples are:

- The researchers believe that it is not in your best interest to stay in the study.
- You become ineligible to participate.
- Your condition changes and you need treatment that is not allowed while you are taking part in the study.
- You do not follow instructions from the researchers.
- The study is suspended or canceled.

IRBMED standard informed consent template (working version)

Approved 4/10/2024
Blue box instructions revised 8/21/2024
DO NOT REMOVE THIS FIELD—IRBMED USE ONLY

Consent Subtitle: \_\_\_Aim 3\_\_\_\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_

#### 8. FINANCIAL INFORMATION

#### 8.1 Who will pay for the costs of the study? Will I or my health plan be billed for any costs of the study?

The study will pay for research-related items or services that are provided only because you are in the study. If you get a bill you think is wrong, call the researcher's telephone number listed in Section 10.1.

By signing this form, you do not give up your right to seek payment if you are harmed because of being in this study.

#### 8.2 Will I be paid or given anything for taking part in this study?

No. You will not be paid for taking part in this study.

#### 8.3 Who could profit or financially benefit from the study results?

No person or organization can profit or financially benefit from the outcome of the study.

The University of Michigan is receiving payments from the Agency for Healthcare Research and Quality to support the activities that are required to conduct the study.

Research can lead to new discoveries, such as new tests, drugs, or devices. Researchers, their organizations, and other entities, including companies, may potentially benefit from the use of the data or discoveries. You will not have rights to these discoveries or any proceeds from them.

# 9. CONFIDENTIALITY OF PARTICIPANT RECORDS AND AUTHORIZATION TO RELEASE YOUR PROTECTED HEALTH INFORMATION

The information below describes how the confidentiality of your research records will be protected in this study, and any sub-studies described in this document.

#### 9.1 How will the researchers protect my information?

Your participation will occur at Michigan Medicine. Your data will be kept confidential, to the extent permitted by applicable laws, in the following manner:

- Your name will not be used in any reports about the study
- You will be identified only by a study code
- Your identifying information will be kept secure

Despite these protections, some study data may contain information that could be used (perhaps in combination with other information) to identify you (e.g., initials, date of birth).

This trial will be registered and may report results on www.ClinicalTrials.gov, a publicly available registry of clinical trials. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

# 9.2 What protected health information (PHI) about me could be seen by the researchers or by other people? Why? Who might see it?

Signing this form gives the researchers your permission to obtain, use, and share information about you for this study, and is required for you to take part in the study.

IRBMED standard informed consent template (working version)

Approved 4/10/2024
Blue box instructions revised 8/21/2024
DO NOT REMOVE THIS FIELD—IRBMED USE ONLY

Consent Subtitle: \_\_\_Aim 3\_\_\_\_\_\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_\_\_\_

Medical information and billing records are protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA). This type of information is called protected health information (PHI). PHI about you may be obtained from any hospital, doctor, and other health care provider involved in your care, including:

- Hospital/doctor's office records, including test results (X-rays, blood tests, urine tests, etc.)
- All records relating to your condition, the treatment you have received, and your response to the treatment
- Demographic information
- Personal identifiers

There are many reasons why information about you may be used or seen by the researchers or others during or after this study. Examples include:

- The researchers may need the information to make sure you can take part in the study.
- The researchers may need the information to check your test results or look for side effects.
- University, Food and Drug Administration (FDA) and/or other government officials, auditors, and/or the IRB may need the information to make sure that the study is done in a safe and proper manner and for quality improvement purposes.
- Study sponsors or funders, or safety monitors or committees, may need the information to:
  - Make sure the study is done safely and properly
  - Learn more about side effects
  - Analyze the results of the study
- Insurance companies or other organizations may need the information to pay your medical bills or other costs of your participation in the study.
- The researchers may need to use the information to create a databank of information about your condition or its treatment.
- Information about your study participation may be included in your regular Michigan Medicine medical record
- Federal or State law may require the study team to give information to government agencies. For example, to prevent harm to you or others, or for public health reasons.

The results of this study could be published in an article, but would not include any information that would let others know who you are.

#### 9.3 What happens to information about me after the study is over or if I cancel my permission to use my PHI?

As a rule, the researchers will not continue to use or disclose information about you, but will keep it secure until it is destroyed. Sometimes, it may be necessary for information about you to continue to be used or disclosed, even after you have canceled your permission or the study is over.

Examples of reasons for this include:

• To avoid losing study results that have already included your information

| | IRBMED standard informed consent template (working version) |
|---|-------------------------------------------------------------|
| | Approved 4/10/2024 |
| | Blue box instructions revised 8/21/2024 |
| E | DO NOT REMOVE THIS FIELD—IRBMED USE ONLY |

Consent Subtitle: \_\_\_Aim 3\_ Consent Version: \_\_\_v1\_5Oct2024\_\_\_\_\_

- To provide limited information for research, education, or other activities. (This information would not include your name, social security number, or anything else that could let others know who you are.)
- To help University and government officials make sure that the study was conducted properly

If your information is kept within the University of Michigan Health System, it is protected by the Health System's privacy policies. For more information about these policies, ask for a copy of the University of Michigan "Notice of Privacy Practices". This information is also available on the web at

http://www.uofmhealth.org/patient+and+visitor+guide/hipaa. Note that once your information has been shared with others as described under Question 9.2, it may no longer be protected by the privacy regulations of the federal Health Insurance Portability and Accountability Act of 1996 (HIPAA).

#### 9.4 When does my permission to use my PHI expire?

Your permission does not expire unless you cancel it. You may cancel your permission at any time by writing to the researchers listed in Section 10 "Contact Information" (below). If you withdraw your permission, you may no longer be eligible to participate in this study.

#### 10. CONTACT INFORMATION

#### 10.1 Who can I contact about this study?

Please contact the researchers listed below to:

- Obtain more information about the study
- Ask a question about the study procedures or treatments
- Talk about study-related costs to you or your health plan
- Report an illness, injury, or other problem (you may also need to tell your regular doctors)
- Leave the study before it is finished
- Express a concern about the study

Principal Investigator: Manjunath (Amit) Pai, PharmD

Mailing Address: College of Pharmacy, 428 Church St., Rm 2568

Ann Arbor, MI 48109-2026

Telephone: 734.647-0006

Study Coordinator: June A Sullivan , MBA Mailing Address: Med Sci I, Room 3317

Ann Arbor, MI 48109-2026

Telephone: 734.615-3488

# You may also express a question or concern about a study by contacting the Institutional Review Board listed below:

University of Michigan Medical School Institutional Review Board (IRBMED) 2800 Plymouth Road

Building 520, Room 3214 Ann Arbor, MI 48109-2800

Telephone: 734-763-4768 (For International Studies, include the appropriate calling codes.)

IRBMED standard informed consent template
(working version)
Approved 4/10/2024
Blue box instructions revised 8/21/2024
DO NOT REMOVE THIS FIELD—IRBMED USE ONLY

Fax: 734-763-1234

e-mail: irbmed@umich.edu

If you are concerned about a possible violation of your privacy or concerned about a study you may contact the University of Michigan Health System Compliance Help Line at 1-866-990-0111.

When you call or write about a concern, please provide as much information as possible, including the name of the researcher, the IRBMED number (at the top of this form), and details about the problem. This will help University officials to look into your concern. When reporting a concern, you do not have to give your name unless you want to.

#### 11. RECORD OF INFORMATION PROVIDED

#### 11.1 What documents will be given to me?

You will receive a copy of the signed and dated informed consent document.

Your signature in the next section means that you have received a copy of the following document(s):

• This "Consent to be Part of a Research Study" document. (Note: In addition to the copy you receive, copies of this document will be stored in a separate confidential research file and may be entered into your regular University of Michigan medical record.)

# 12. STORAGE, USE, AND SHARING OF SPECIMENS AND INFORMATION COLLECTED OR GENERATED IN THE STUDY DESCRIBED ABOVE

# 12.1 What is meant by the storage, future research use, and sharing of study participants' medical information and leftover samples (sometimes referred to as biospecimens) taken from me?

Individual researchers, the University of Michigan, and companies that design and sponsor studies often want to keep subjects' medical information and leftover samples such as blood, tissue, saliva, and cells to use in future research. These future research uses take different basic forms, which are described below. The medical information and leftover samples may also be shared with other researchers so that they can use it in their studies.

The purpose of storing, using, and sharing participants' medical information and leftover samples is to promote more research that might lead to useful medical discoveries.

In some cases, researchers need your consent to store, use, and share your medical information and leftover samples; in other cases, they can store, use and/or share it without your consent. Whether or not researchers need your consent depends on if the stored information and samples would still be identifiable as yours or whether the researchers would first remove all information connecting them back to you.

#### 12.2 Types of storage, future research use, and sharing in this study

We would also like your permission to keep some of your identifiable blood, fat, and appendix tissue samples and medical information collected in the main study, so that it may be studied it in future research. The future research may be similar to this study or may be completely different.

You can take part in the main study even if you decide not to let us keep your identifiable blood, fat, and appendix tissue samples and medical information for future research.

If you give us your permission, we will use your identifiable blood, fat, and appendix tissue samples and medical information for future research. Even if you give us permission now to keep some of your identifiable blood, fat, and

| IRBMED standard informed consent template (working version) |
|-------------------------------------------------------------|
| Approved 4/10/2024 |
| Blue box instructions revised 8/21/2024 |
| DO NOT REMOVE THIS FIELD—IRBMED USE ONLY |

appendix tissue samples and study information collected in the study, you can change your mind later and ask us to destroy it. If you do change your mind, we will attempt to get your information and biospecimens back from the other researchers we've shared them with. However, there may be times we cannot. For example, if we are unable to tell which information and biospecimens came from you, we will not be able to get them back. Additionally, any information that has been added to your medical record cannot be deleted. Also, keep in mind that once we have analyzed your blood, fat, and appendix tissue samples we may not be able to take the information out of our research study.

We may share your blood, fat, and appendix tissue samples and medical information with other researchers, so that they can use it in their research. Their research may be similar to this study or may be completely different. Once we have shared your blood, fat, and appendix tissue samples and medical information with other researchers, we will not be able to get it back.

Although we will do our best to protect your information and specimens, both during storage and when sharing them with others, it's possible that someone may be able to identify you from them. It's also possible that unauthorized people might gain access your information and/or specimens. To try to minimize both of these risks, we will assign your information and specimens a random code before sharing them with other researchers. Dr. Manjunath (Amit) Pai will securely store the code key that links your coded information and specimens to you. Future use of your identifiable data and/or specimens will be conducted in compliance with applicable regulatory requirements.

You will not find out the results or benefit directly from future research on your blood, fat, and appendix tissue samples. Sharing your information and specimens may contribute to research that helps others in the future

#### 13. SIGNATURES

| | Sig-A |
|---|---|
| Consent/Assent to Participate in the Research Study | |
| I understand the information printed on this form. I have discussed this study, its risks and potential ber and my other choices with [NAME OF STUDY TEAM MEMBER OBTAINING CONSENT] | - |
| My questions so far have been answered. I understand that if I have more questions or concerns about study or my participation as a research subject, I may contact one of the people listed in Section 10 (abounderstand that I will receive a copy of this form at the time I sign it and later upon request. I understand my ability to consent or assent for myself changes, either I or my legal representative may be asked to reconsent prior to my continued participation in this study. | ove). I<br>nd that if |
| Print Legal Name: | |
| Signature: | |
| Date of Signature (mm/dd/yy): | |

IRBMED standard informed consent template (working version)

Approved 4/10/2024
Blue box instructions revised 8/21/2024

DO NOT REMOVE THIS FIELD—IRBMED USE ONLY

| Consent/Assent to Collect for Unspecified Future Research This project involves the option to allow the study team to keep your identifiable specimens/data for use in future research. I understand that it is my choice whether or not to allow future use of my specimens. I understand that if my ability to consent or assent for myself changes, either I or my legal representative may be asked to re-consent prior to my continued participation in this study. Yes, I agree to let the researchers keep my specimens for future research (signature required below). No, I do not agree to let the researchers keep my specimens for future research (no signature). |
|---|
| Print Legal Name: |
| Signature: |
| Date of Signature (mm/dd/yy): |
| Sig-G |
| Principal Investigator or Designee I have provided this participant and/or his/her legally authorized representative(s) with information about this study that I believe to be accurate and complete. The participant and/or his/her legally authorized representative(s) indicated that he or she understands the nature of the study, including risks and benefits of participating. |
| Printed Legal Name: |
| Title: |
| Signature: |
| Date of Signature (mm/dd/yy): |

IRBMED standard informed consent template (working version)

Approved 4/10/2024
Blue box instructions revised 8/21/2024
DO NOT REMOVE THIS FIELD—IRBMED USE ONLY